CLINICAL TRIAL: NCT03127774
Title: Phase II Trial of Surgical Resection and Heated Intraperitoneal Peritoneal Chemotherapy (HIPEC) for Adrenocortical Carcinoma
Brief Title: Surgery and Heated Intraperitoneal Chemotherapy for Adrenocortical Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Kazuki Sugahara, Assistant Professor of Surgery, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ9194
Record Dates: First submitted 2017-04-02; First posted 2017-04-25 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Adrenocortical Carcinoma; Peritoneal Carcinomatosis
Keywords: Cisplatin; Heated Cisplatin
MeSH Terms: conditions — Adrenocortical Carcinoma; Peritoneal Neoplasms | interventions — Cisplatin; sodium thiosulfate; Cytoreduction Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Patients who are successfully debulked will undergo heated intraperitoneal chemotherapy with cisplatin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surgery with HIPEC (Experimental): Cytoreductive surgery followed by HIPEC with cisplatin and sodium thiosulfate
  Interventions: Drug: Cisplatin; Drug: Sodium thiosulfate; Procedure: Cytoreductive surgery

INTERVENTIONS:
Drug: Cisplatin — Route of administration: Intraperitoneal for tumor treatment. Dose of 250 mg/m2
  Drug 1 of the hyperthermic intraperitoneal chemotherapy (HIPEC)
  Other Names: Platinol
Drug: Sodium thiosulfate — Route of administration: Intravenous Loading dose of 7.5 gm/m2 over 20 minutes followed by 2.13 gm/m2/hr for 12 hours
  Drug 2 given intravenously during hyperthermic intraperitoneal chemotherapy (HIPEC)
  Other Names: Sodium thiosulfate injection
Procedure: Cytoreductive surgery — Standard of care: Surgical procedure used to remove tumors from patients with peritoneal tumors.
  Other Names: Cytoreductive debulking surgery

SUMMARY:
Objectives:

- To determine intraperitoneal (IP) progression free survival after optimal debulking and heated intraperitoneal chemotherapy (HIPEC) with cisplatin in patients with IP spread of adrenocortical cancer.

- Determine morbidity of this procedure in this patient population.

- Determine the impact of surgery and HIPEC on quality of life (QOL) and hormone excess.

- Examine patterns of recurrence (local versus systemic).

- Determine overall survival after optimal debulking and HIPEC in patients with IP spread of adrenocortical cancer.

DETAILED DESCRIPTION:
Adrenocortical carcinoma (ACC) is a rare tumor with an overall 5-year mortality rate of 75 - 90% and an average survival from the time of diagnosis of 14.5 months. The treatment of choice for a localized primary or recurrent tumor is surgical resection of all visible tumor and involved organs. For unresectable metastatic or recurrent disease, mitotane, aminoglutethimide, metapyrone, and ketoconazole are used. This would be the standard of care alternative treatment.

Cisplatin is one of the most effective chemotherapeutic agents for ACC. Phase I and II trials using heated intraperitoneal (IP) chemotherapy with cisplatin have been conducted in other tumors that spread primarily to the peritoneal lining of the abdomen. Synergy has been demonstrated for cisplatin and hyperthermia. The purpose of this trial is to determine if an surgical approach with intraperitoneal administration of heated cisplatin when tumor volume is minimal, can impact and improve on progression free survival.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically proven ACC with the majority of disease confined to the peritoneal cavity and resectable or amenable to radiofrequency ablation
* Disease evaluable by CT or Positron Emission Tomography (PET) imaging
* All disease should be deemed resectable based on imaging studies e.g.:

  * Hepatic metastases (unilateral or bilateral less than or equal to 5 lesions, less than or equal to 15 cm total diameter)
  * Note: Hepatic lesions must be amenable to complete resection
  * Primary peritoneal metastases (small disease load less than or equal to P2 disease) without massive ascites or intestinal obstruction
  * Lung metastases (less than or equal to 3 unilateral/bilateral, 9 cm total diameter)
  * Note: lung lesions must be amenable to complete resection
  * Note: Patients with both pulmonary and hepatic metastases will be enrolled at the discretion of the PI
  * Note: In situations where resection to Completeness of Cytoreduction Score (CC) 0 or 1 is uncertain, patients may undergo diagnostic laparoscopy prior to enrollment to determine feasibility of resection.
* Greater than or equal to 18 years of age
* Able to understand and sign the Informed Consent Document
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) less than or equal to 2
* Life expectancy of greater than three months
* Patients of both genders must be willing to practice birth control during and for four months after receiving chemotherapy
* Hematology:

  * Absolute neutrophil count greater than 1500/mm^3 without the support of Filgrastim.
  * Platelet count greater than 75,000/mm^3.
  * Hemoglobin greater than 8.0 g/dl.
* Chemistry:

  * Serum creatinine less than or equal to 1.5 mg/dl unless the measured creatinine clearance is greater than 60 mL/min/1.73 m2
  * serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within 5 times the upper limit of normal and a total serum bilirubin of less than 3 times the upper limit of normal, both of which define the upper limit of grade 2 treatment related toxicities.
  * Prothrombin time (PT) within 2 seconds of the upper limit of normal (INR less than or equal to 1.8)
* Recovered from any toxicity to grade 2 or less from all prior chemotherapy, immunotherapy or radiotherapy and be at least 30 days past the date of their last treatment with the exception of mitotane which may be continued.
* Able to understand their disease and the exploratory nature of combining surgery and HIPEC for this histology.

EXCLUSION CRITERIA

* Concomitant medical problems that would place the patient at unacceptable risk for a major surgical procedure.
* History of congestive heart failure and/or an left ventricular ejection fraction (LVEF) less than 40%

Note: Patients at increased risk for coronary artery disease or cardiac dysfunction (e.g., greater than 65yo, diabetes, history of hypertension, elevated LDL, first degree relative with coronary artery disease) will undergo full cardiac evaluation and will not be eligible if they demonstrate significant irreversible ischemia on stress thallium or an ejection fraction less than 40%.

- Significant chronic obstructive pulmonary disease (COPD) or other chronic pulmonary restrictive disease with pulmonary function test (PFT) indicating an forced expiratory volume at one second (FEV1) less than 50% or a diffusing capacity of lung for carbon monoxide (DLCO) less than 40% predicted for age.

Note: Patients who have shortness of breath with minimal exertion or who are at risk for pulmonary disease (e.g., chronic smokers) will undergo pulmonary function testing and will not be eligible if their FEV1 is less than 50% of expected.

* Grade 2 or greater neuropathy
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the chemotherapy on the fetus or infant.
* Brain metastases or a history of brain metastases
* Childs B or C cirrhosis
* Evidence of severe portal hypertension by history, endoscopy, or radiologic studies

Note: Any diagnosis of portal hypertension or clinical stigmata of such including but not limited to gastric or esophageal varices, umbilical vein varices or telangiectasias.

* Weight less than 30 kg
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 5 years
  The length of time after optimal debulking and heated intraperitoneal chemotherapy that a patient lives before there is clinical evidence of recurrent adrenocortical cancer.

SECONDARY OUTCOMES:
Morbidity Rate | Up to 5 years
  The frequency of post-operative complications.
Quality of Life (QOL) Score | Up to 5 years
  This measures the impact of surgery and HIPEC on quality of life.
Overall Survival | Up to 5 years
  The length of time people are alive after surgery and HIPEC for adrenocortical cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuki Sugahara, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No